CLINICAL TRIAL: NCT05451901
Title: Immediate Necrosectomy vs. Step-up Approach After EUS-guided Drainage of Walled-off Necrosis: a Multicenter Randomized Controlled Trial (WONDER-01)
Brief Title: Immediate Necrosectomy vs. Step-up Approach for Walled-off Necrosis
Acronym: WONDER-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tokyo University (Other)
Responsible Party: Principal Investigator, Yousuke Nakai, Associate professor, Department of Endoscopy and Endoscopic Surgery, The University of Tokyo Hospital, Tokyo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021005P; jRCT1032220055 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2022-07-03; First posted 2022-07-11 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Pancreatic Fluid Collection; Walled-off Necrosis; Pancreatitis, Acute Necrotizing; Pancreatic Pseudocyst
Keywords: Endosonography; Drainage; Stents; Endoscopic necrosectomy; Step-up approach
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing; Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate necrosectomy (Experimental): Endoscopic necrosectomy will be conducted in the same session of EUS-guided drainage (or at least within 72 hours of randomization) and be repeated until clinical success.
  Interventions: Procedure: Immediate necrosectomy
- Step-up approach (Active Comparator): Step-up treatment will be conducted if a patient's condition does not improve after EUS-guided drainage. The step-up approach includes increasing the number of stents, adding another EUS-guided drainage, and performing percutaneous drainage after 72-96 hours of the initial drainage. Endoscopic necrosectomy is considered when clinical improvement is not observed even after two times of step-up treatment.
  Interventions: Procedure: Step-up approach

INTERVENTIONS:
Procedure: Immediate necrosectomy — Endoscopic ultrasonography (EUS)-guided drainage will be conducted within 72 hours from randomization. A convex-type echoendoscope is advanced to the stomach or duodenum, and the walled-off necrosis (WON) is visualized and punctured under EUS guidance. A lumen-apposing metal stent (LAMS), such as Hot AXIOS system (Boston Scientific Japan, Tokyo, Japan), is recommended for the initial EUS-guided drainage.
  For the immediate necrosectomy group, endoscopic necrosectomy (EN) will be performed in the same session of EUS-guided drainage using a gastroscope. The endoscope is inserted into the WON cavity through the LAMS, and necrotic tissue is removed using biopsy forceps, snare, or basket catheter. The EN procedures will be repeated until clinical improvement.
  Arms: Immediate necrosectomy
Procedure: Step-up approach — Endoscopic ultrasonography (EUS)-guided drainage will be conducted within 72 hours from randomization. A convex-type echoendoscope is advanced to the stomach or duodenum, and the walled-off necrosis (WON) is visualized and punctured under EUS guidance. A lumen-apposing metal stent (LAMS), such as Hot AXIOS system (Boston Scientific Japan, Tokyo, Japan), is recommended for the initial EUS-guided drainage.
  For the step-up approach group, an additional interventional procedure will be withheld for 72-96 hours after initial EUS-guided drainage. In cases without clinical improvement after 72-96 hours, additional drainage will be permitted, which includes increasing the number of stents, additional EUS-guided drainage, and performing percutaneous drainage (step-up treatment). Insufficient improvement even after two times of step-up treatment allows subsequent endoscopic necrosectomy (EN).
  Arms: Step-up approach

SUMMARY:
Walled-off necrosis (WON) is a pancreatic fluid collection, which contains necrotic tissue after four weeks of the onset of acute pancreatitis. Interventions are required to manage patients with infected WON, for which endoscopic ultrasonography (EUS)-guided drainage has become a first-line treatment modality. For patients who are refractory to EUS-guided drainage, the step-up treatment including endoscopic necrosectomy (EN) and/or additional drainage is considered to subside the infection. Recent evidence suggests that EN immediately after EUS-guided drainage may shorten treatment duration without increasing adverse events. In this randomized trial, the investigators will compare treatment duration between EN immediately after EUS-guided drainage versus the step-up approach in patients with symptomatic WON.

DETAILED DESCRIPTION:
Pancreatic fluid collection is a late complication of severe acute pancreatitis. According to the revised Atlanta classification, walled-off necrosis (WON) is defined as an encapsulated collection of necrotic tissue that is observed after four weeks of the onset of acute pancreatitis. Infected WON is associated with high morbidity and mortality; therefore, an appropriate treatment, including antibiotics and drainage, is mandatory. With the development of endoscopic equipment, endoscopic ultrasonography (EUS)-guided drainage has become a first-line treatment modality for infected WON. For patients who are refractory to EUS-guided drainage, endoscopic necrosectomy (EN) is a treatment option to facilitate direct removal of infected necrotic tissue within the WON. However, due to potentially lethal adverse events of EN, such as bleeding, perforation, and peritonitis, EN is usually withheld for several days after EUS-guided drainage. This strategy is known as "the step-up approach." Recently, with the accumulated evidence supporting the safety of EN, especially with the use of a dedicated lumen-apposing metal stent, it has been reported that EN immediately after EUS-guided drainage can shorten the treatment duration without increasing adverse events. Given these lines of evidence, the investigators hypothesized that immediate EN following EUS-guided drainage of WON might shorten time to clinical success compared to the step-up approach. To examine this hypothesis, the investigators planned to conduct a multicenter randomized controlled trial comparing treatment duration between EN immediately after EUS-guided drainage versus the step-up approach in patients with symptomatic WON.

ELIGIBILITY:
Inclusion Criteria:

* Patients with WON defined according to the revised Atlanta classification
* The longest diameter of WON is 4 cm or larger
* Patients with at least one out of the following conditions; signs of infection, gastrointestinal symptoms, abdominal symptoms, obstructive jaundice
* Patients who need drainage for WON
* Age of 18 years or older
* Patients or their representatives provide informed consent
* Patients who visit or are hospitalized at the participating institutions

Exclusion Criteria:

* WON inaccessible by EUS-guided approach
* AXIOS stent has already been placed into the WON prior to the enrollment
* Severe coagulopathy; Platelet count < 50,000/mm3 or prothrombin time international normalized ratio (PT-INR) >1.5
* Patients on antithrombotic agents which cannot be managed according to the "guideline for gastroenterological endoscopy in patients undergoing antithrombotic treatment (Dig Endosc. 2014 Jan;26(1):1-14.)"
* Patients who cannot tolerate endoscopic procedures
* Pregnant women
* Patients considered inappropriate for inclusion by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2031-04-11 (Estimated)

PRIMARY OUTCOMES:
Time to clinical success from randomization | Six months
  Clinical success is defined as 1) a decrease in the WON size to 3 cm or less and 2) an improvement of more than two out of the three following inflammatory markers; body temperature, white blood cell count, and C-reactive protein.

SECONDARY OUTCOMES:
Adverse events | Five years
  All procedure-related adverse events including bleeding, perforation, peritonitis, etc.
Mortality | Five years
  Mortality from any cause
Technical success rate of initial EUS-PCD (Endoscopic ultrasonography-guided pseudocyst drainage) | One day
  Successful placement of EUS-guided drainage including a lumen-apposing metal stent and plastic stents
Incidence of biliary and gastrointestinal stricture | Five years
  Inflammatory-induced obstruction of bile duct and gastrointestinal tract
Number and time of interventions | Six months
  Total number of interventions and total procedure time
Indwelling time of endoscopic and percutaneous drainage | Six months
  Indwelling period of stents and drainage tube
Success rate and operation time of surgical procedures | Six months
  Success rate of surgeries associated with WON and total operation time
Hospital stay and ICU stay | Six months
  Total hospitalization days and total ICU stay
Duration of antibiotics administration | Six months
  Total administration days of antibiotics
Cost of interventions and hospital stay | Six months
  Total cost of interventions and total cost of hospitalization
Recurrence of WON | Five years
  Incidence of recurrence of WON
Time to recurrence of WON | Five years
  Time from clinical success to recurrence of WON
Treatment duration of recurrent WON | Five years
  Total treatment period for recurrent WON
New onset of pseudocyst | Five years
  Incidence of new-onset pancreatic pseudocyst
Treatment duration of new onset pseudocyst | Five years
  Total treatment period for new-onset pancreatic pseudocyst
Incidence of new onset diabetes, clinical symptoms of pancreatic exocrine insufficiency, and pancreatic cancer | Five years
  New-onset diabetes mellitus, pancreatic cancer, and clinical symptoms associated with pancreatic exocrine insufficiency, such as steatorrhea , constipation, diarrhea, maldigestion, flatulence, and tenesmus
The presence and timing of medications for pancreatic exocrine insufficiency | Five years
  The start of medications for pancreatic exocrine insufficiency and the date
The presence and timing of sarcopenia | Five years
  The presence of sarcopenia and the date of diagnosis
Morphological change of pancreas | Five years
  Change in the morphology and the volume of pancreas

CONTACTS AND LOCATIONS:
Overall Officials: Yousuke Nakai, Principal Investigator — Department of Endoscopy and Endoscopic Surgery, Graduate School of Medicine, The University of Tokyo
Locations (21):
- Japan (21):
  - Department of Gastroenterology, The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - Department of Gastroenterology, Graduate School of Medicine, Juntendo University, Bunkyō-Ku, Tokyo
  - Department of Gastroenterology, Aichi Medical University, Aichi
  - Department of Gastroenterology, Graduate School of Medicine, Chiba University, Chiba
  - Department of Gastroenterology, Gifu Municipal Hospital, Gifu
  - Department of Gastroenterology, Gifu Prefectural General Medical Center, Gifu
  - First Department of Internal Medicine, Gifu University Hospital, Gifu
  - Division of Gastroenterology and Hepatobiliary and Pancreatic Diseases, Department of Internal Medicine, Hyogo Medical University, Hyōgo
  - Department of Gastroenterology and Neurology, Faculty of Medicine, Kagawa University, Kagawa
  - Digestive and Lifestyle Diseases, Kagoshima University Graduate School of Medical and Dental Sciences, Kagoshima
  - Department of Gastroenterology, Kameda Medical Center, Kamogawa
  - Department of Gastroenterological Endoscopy, Kanazawa Medical University, Kanazawa
  - Department of Gastroenterology and Hepatology, Saitama Medical Center, Saitama Medical University, Kawagoe
  - Department of Gastroenterology, Teikyo University Mizonokuchi Hospital, Kawasaki
  - Division of Gastroenterology, Department of Internal Medicine, Kobe University Graduate School of Medicine, Kobe
  - Department of Gastroenterology, Yuuai Medical Center, Okinawa
  - 2nd Department of Internal Medicine, Osaka Medical College, Osaka
  - Department of Gastroenterology and Hepatology, Kindai University Faculty of Medicine, Ōsaka-sayama
  - Department of Gastroenterology and Hepatology, Hokkaido University Hospital, Sapporo
  - Division of Gastroenterology and Hepatology, Department of Medicine, Nihon University School of Medicine, Tokyo
  - Third Department of Internal Medicine, University of Toyama, Toyama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Derived] Sato T, Saito T, Takenaka M, Iwashita T, Shiomi H, Fujisawa T, Hayashi N, Iwata K, Maruta A, Mukai T, Masuda A, Matsubara S, Hamada T, Inoue T, Ohyama H, Kuwatani M, Kamada H, Hashimoto S, Shiratori T, Yamada R, Kogure H, Ogura T, Nakahara K, Doi S, Chinen K, Isayama H, Yasuda I, Nakai Y; WONDERFUL study group in Japan, collaborators. WONDER-01: immediate necrosectomy vs. drainage-oriented step-up approach after endoscopic ultrasound-guided drainage of walled-off necrosis-study protocol for a multicentre randomised controlled trial. Trials. 2023 May 24;24(1):352. doi: 10.1186/s13063-023-07377-y. PMID 37226252